CLINICAL TRIAL: NCT00958269
Title: A Randomized, Double-Blind, Placebo- and Sitagliptin-Controlled, Multi-Center Study to Evaluate Safety and Efficacy of Dutogliptin in Type 2 Diabetes Mellitus Subjects With Moderate and Severe Renal Impairment Including Subjects on Hemodialysis
Brief Title: Study to Evaluate Safety and Efficacy of Dutogliptin in Type 2 Diabetes Mellitus Subjects With Moderate and Severe Renal Impairment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Technical/operational issues
Sponsor: Phenomix (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Hans-Peter Guler, MD, Phenomix Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHX1149-PROT306
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Type 2 Diabetes Mellitus; Renal Impairment
Keywords: diabetes; DPP4 inhibitor; dutogliptin; PHX1149
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency; Diabetes Mellitus | interventions — dutogliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- dutogliptin (double-blind, placebo-controlled period) (Experimental): weeks 1-26
  Interventions: Drug: dutogliptin
- dutogliptin (single-blind, active-controlled period) (Experimental): weeks 27-52
  Interventions: Drug: dutogliptin
- placebo (double-blind, placebo-controlled period) (Placebo Comparator): weeks 1-26
  Interventions: Drug: placebo
- placebo (single-blind, active-controlled period) (Placebo Comparator): weeks 27-52
  Interventions: Drug: placebo
- sitagliptin (single-blind, active-controlled period) (Active Comparator): weeks 27-52
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: dutogliptin — 100 mg QD
  Arms: dutogliptin (double-blind, placebo-controlled period); dutogliptin (single-blind, active-controlled period)
Drug: dutogliptin — 200 mg QD
  Arms: dutogliptin (double-blind, placebo-controlled period); dutogliptin (single-blind, active-controlled period)
Drug: placebo
  Arms: placebo (double-blind, placebo-controlled period); placebo (single-blind, active-controlled period)
Drug: sitagliptin — 25 mg QD
  Arms: sitagliptin (single-blind, active-controlled period)
Drug: sitagliptin — 50 mg QD
  Arms: sitagliptin (single-blind, active-controlled period)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of dutogliptin in Type 2 diabetic subjects with moderate or severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Renal impairment (moderate and severe)
* Currently on stable doses of background medication of SU, TZD, acarbose, meglitinide, insulin or any combination thereof, or on no antidiabetic drugs at all
* HbA1c 7.0% - 10.5%, inclusive
* Male or female subjects between the ages of 18 and 85 years, inclusive.

Exclusion Criteria:

* Type 1 diabetes mellitus or history of diabetic ketoacidosis, mature onset diabetes of the young (MODY)
* Kidney transplant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of dutogliptin as assessed by analysis of AEs/SAEs, laboratory data, vital signs, and ECGs | Day 1 through day 182 (end of the 26-week, double-blind, placebo-controlled period) and through Day 364 (end of the 26-week, sitagliptin-controlled period of the study)

SECONDARY OUTCOMES:
Change of HbA1c | Day 1 to Day 182
Change of fasting plasma glucose | Day 1 to Day 182
Plasma dutogliptin levels | Days 1, 198 and 182
Per cent ex vivo DPP4 inhibition after drug dosing | Days 1, 98, and 182

CONTACTS AND LOCATIONS:
Locations (43):
- United States (23):
  - Phenomix Investigational Site 115, Tempe, Arizona
  - Phenomix Investigational Site 121, Long Beach, California
  - Phenomix Investigational Site 110, Lynwood, California
  - Phenomix Investigational Site 118, Lynwood, California
  - Phenomix Investigational Site 119, Orange, California
  - Phenomix Investigational Site 109, Palm Springs, California
  - Phenomix Investigational Site 122, Whittier, California
  - Phenomix Investigational Site 112, Lauderdale Lakes, Florida
  - Phenomix Investigational Site 104, Ocala, Florida
  - Phenomix Investigational Site 116, Pembroke Pines, Florida
  - Phenomix Investigational Site 101, Augusta, Georgia
  - Phenomix Investigational Site 117, Honolulu, Hawaii
  - Phenomix Investigational Site 102, Baton Rouge, Louisiana
  - Phenomix Investigational Site 100, Rockville, Maryland
  - Phenomix Investigational Site 125, Rockville, Maryland
  - Phenomix Investigational Site 114, Springfield Gardens, New York
  - Phenomix Investigational Site 120, Winston-Salem, North Carolina
  - Phenomix Investigational Site 107, Columbia, South Carolina
  - Phenomix Investigational Site 111, Nashville, Tennessee
  - Phenomix Investigational Site 103, Fort Worth, Texas
  - Phenomix Investigational Site 106, Houston, Texas
  - Phenomix Investigational Site 108, San Antonio, Texas
  - Phenomix Investigational Site 113, Alexandria, Virginia
- Russia (13):
  - Phenomix Investigational Site 208, Kemerovo
  - Phenomix Investigational Site 203, Moscow
  - Phenomix Investigational Site 204, Moscow
  - Phenomix Investigational Site 209, Moscow
  - Phenomix Investigational Site 211, Moscow
  - Phenomix Investigational Site 205, Novosibirsk
  - Phenomix Investigational Site 207, Perm
  - Phenomix Investigational Site 206, Petrozavodsk
  - Phenomix Investigational Site 200, Saint Petersburg
  - Phenomix Investigational Site 201, Saint Petersburg
  - Phenomix Investigational Site 210, Saint Petersburg
  - Phenomix Investigational Site 212, Saint Petersburg
  - Phenomix Investigational Site 213, Saint Petersburg
- Ukraine (7):
  - Phenomix Investigational Site 304, Chernivtsi
  - Phenomix Investigational Site 300, Kyiv
  - Phenomix Investigational Site 301, Kyiv
  - Phenomix Investigational Site 306, Kyiv
  - Phenomix Investigational Site 302, Odesa
  - Phenomix Investigational Site 303, Vinnytsa
  - Phenomix Investigational Site 307, Zaporizhzhya